The University of Michigan PCOS Intervention Using Nutritional Ketosis

NCT03987854

10/31/2019

# The PINK Study (PCOS Intervention using Nutritional Ketosis): Diet and lifestyle management for women with polycystic ovary syndrome

Principal Investigator
Laura Saslow, PhD

## **Proposal**

# 1.0 Objective and Specific Aim/Hypothesis for this IRB application:

The goal of this proposed research is to pilot our existing LCD intervention for type 2 diabetes to use in overweight or women with PCOS.

Aims: Test the feasibility, acceptability, and preliminary efficacy of the intervention. We will randomize 30 overweight or obese women with PCOS to the 4-month intervention. Outcome measures include:

- **intervention feasibility** (recruitment and retention);
- acceptability (satisfaction with the intervention); and
- **preliminary efficacy** as determined by our primary outcome (body weight), as well as and other measures (including glycemic control, insulin resistance, lipids, testosterone, inflammation, and quality of life).

Information gained from this study will be used to finalize the intervention and prepare our team to propose a larger-scale, longitudinal, randomized controlled trial. Ideally, this follow-up trial would also examine long-term adherence and other health implications, including clinical complications. This later research would be appropriate for NIDDK (where Dr. Saslow already has a K01 with Dr. Aikens as mentor).

# 2.0 Background Information: SIGNIFICANCE

Polycystic ovary syndrome (PCOS) is a common and costly disorder. Polycystic ovary syndrome (PCOS) is the most common endocrine disorder for women of reproductive age [1]. Women with PCOS have a 3-7 times higher risk for type 2 diabetes [2], and obese women with PCOS have an even higher risk of type 2 diabetes [3, 4]. Obesity and PCOS tend to co-occur; about 30-60% of women with PCOS are obese [5] and over 10% of obese women have PCOS [6].

Position statements of the Androgen Excess and PCOS Society call for lifestyle management to be the primary treatment for metabolic complications in women with PCOS [7, 8] and the Endocrine Society's clinical practice guideline calls for diet and lifestyle interventions for all overweight or obese women with PCOS [9]. Weight loss, a critical outcome in diet and lifestyle interventions for women with PCOS, may also improve reproductive and metabolic outcomes: reduce insulin, insulin resistance, and androgen levels; improve ovulatory function and pregnancy and live birth rates; and improve glycemic control [7-12]. While experts largely agree that physical activity should be included in such interventions [13, 14], the ideal diet is still debated, especially whether a lower carbohydrate diet is beneficial [12, 15]. The hyperinsulinemia of PCOS likely contributes to the hyperandrogenism, which is why insulin-sensitizing drugs have been proposed as

therapies for PCOS [16]. Reducing insulin through diet, however, may provide a critical nonpharmacological treatment for overweight or obese women with PCOS [17-21].

# 3.0 Methodology:

Participant recruitment and eligibility. We will contact the pool of potentially eligible participants, based on electronic medical records at the University of Michigan, sending them a letter describing the study, which we will also follow up with a phone call. We will also use flyers posted throughout our institution as well as advertise locally, in our referral areas, on our web site and on a variety of other institutional web sites including https://umhealthresearch.org/ and national websites such as PCOS support groups. We will also promote the study to other physicians and healthcare providers.

*Inclusion criteria:* The most generally agreed upon approach to diagnose PCOS is through the Rotterdam criteria. We will include women in one PCOS subtype, those having these two symptoms:

- Hyperandrogenism (a) If not on current birth control: hyperandrogenism defined as current elevated total testosterone >= 50 ng/dL or free androgen index > 1.5 (ratio of testosterone/SHBG x 100) or severe acne or hirsutism (b) if on current birth control: history from the past 10 years of hyperandrogenism defined as past elevated total testosterone >= 50 ng/dL or free androgen index > 1.5 (ratio of testosterone/SHBG x 100) or severe acne or hirsutism
- oligomenorrhea-anovulation defined as spontaneous intermenstrual periods of ≥ 45 days or a total of ≤ 8 menses per year.

We will include participants who, according to the medical records or their self-report, have an existing PCOS diagnosis, plus the following labs from the past 10 years (either from UM medical records, the medical records they choose to send us, or tests that we order for them at baseline):

- total testosterone < 100 ng/dL (required)</li>
- dehydroepiandrosterone sulfate (DHEAS) < 600 μg/dL (required)</li>
- fasting 17-hydroxyprogesterone (17-OHP) level < 2.0 ng/mL (required)</li>
- hyperprolactinaemia (prolactin < 25ng/ml) (required)</li>
- follicle-stimulating hormone (FSH) levels < 20 mIU/mL (optional)</li>

Participants must also be overweight or obese (BMI 25-50), be 21-40 years old, have regular access to the internet, be able to engage in light physical activity, and willing and able to follow the assigned intervention. Their participation in the trial will need to be approved by their primary care physician or another healthcare provider who functions as their primary care physician, such as an endocrinologist.

Exclusion criteria: a non-English speaker; inability to complete baseline measurements; a substance abuse, mental health, or medical condition that would interfere with participation (such as current chemotherapy); pregnant or planning to get pregnant in the next 6 months; type 1 or type 2 diabetes; baseline aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 times normal; baseline renal disease defined as BUN > 30 mg/dL or serum creatinine >1.4 mg/dL; baseline uncorrected thyroid disease (TSH <0.45 mlU/ML or >4.5 mlU/ML); breastfeeding or less than 6 months post-partum; planned or history of weight loss surgery; vegan or vegetarian; currently enrolled in a weight loss program or other investigative study that might conflict with this research; taking medications known to cause weight gain or loss; taking hypoglycemic medications other than metformin or medications known to affect metabolism; or patients with other etiologies of anovulation and hyperandrogenism, e.g., Cushing's disease, thyroid dysfunction, elevated prolactin levels, sighs of congenital adrenal hyperplasia, organic intra cranial lesion such as a pituitary tumor, or suspected adrenal or ovarian tumor secreting androgens.

After passing preliminary eligibility based on an online screening survey (using an online consent form), we will ask participants to (1) have their primary physician approve their participation in the trial, (2) answer online surveys about self-reported physical and psychological well-being, (3) go to one of more than 20 local locations to get their blood measured, (4) perform a 3-day food diary, and (5) weigh themselves on the bodyweight scale that we will mail them.

At month 4 the steps listed above (2-5) will be repeated. In addition, all enrolled participants will be invited to voluntarily participate in an interview at the end of their 4-month intervention. These interviews will explore their perspectives about the feasibility and acceptability of the intervention, as well as barriers and facilitators of their participation. This interview will take place over the phone with study staff and will last approximately 20-30 minutes. The interview will be recorded, saved onto encrypted devices, and then deleted from the recording device. Interviews will be transcribed and then coded by multiple coders to find common, broad themes. We plan to use Production Transcripts (<a href="https://www.productiontranscripts.com/qualitative-research-transcription/">https://www.productiontranscripts.com/qualitative-research-transcription/</a>) to transcribe all interviews and NVivo software for qualitative coding.

**Intervention**. Participants will be e-mailed links to the coursework every week for 16 weeks. We chose this time frame so as to be able to develop a sufficiently robust intervention for the future larger, longer trial. In addition, as HbA1c can take about 3 months to reflect changes in blood glucose control and participants may take 1 month to fully change their diet to be LCD, 4 months should yield an accurate estimate of the changes in their blood glucose control.

The weekly links will connect participants to: a) a short survey to assess intervention-related behavioral adherence and any health concerns, b) a short embedded video to teach the topics, c) downloadable handouts distributed online to accompany the videos, and d) links to external resources on the web pertaining to the week's information. As some participants prefer not to watch videos, the transcripts of the embedded videos will be provided as well, in an easy-to-read downloadable pdf format.

The lessons will not be delivered synchronously in real time, but will be able to be watched and read whenever is convenient. Participants will be encouraged to complete the lessons in one sitting although they will be able to log into the lesson again at a later point if they would prefer. Lessons will vary in length, but on average they will take about 10 to 30 minutes to complete, including watching the short video and reading the handouts. We will track how often and when participants log into the lessons, thus allowing us to assess engagement with the curriculum.

Some of the intervention topics and approaches are described below:



**Dietary Component: An LCD**. Participants will be encouraged to eat an LCD, the same one Dr. Saslow has recommended in her previous research [22, 23], to reduce carbohydrate intake to between 20-35 non-fiber grams of carbohydrates a day. Participants will be encouraged to eat a normal amount of protein (to keep their protein levels as they were before the intervention began, as long as they were meeting the minimum amount suggested by the Institute of Medicine [24] ) and to derive their remaining calories from fat. Generally, calories will be derived from animal foods, cheeses, eggs, fats, nuts, seeds, and low-carbohydrate vegetables. This intervention was created in consultation with experts in the LCD and has been iterated in six previous trials for adults with prediabetes or type 2 diabetes.

#### **Core Intervention:**

- a) Dietary self-monitoring using a free application. We will ask participants to track their diet using a free online and mobile application, MyFitnessPal (which our participants have found easy to use, has a wide variety of foods in its database, and has over 150 million users). If by the time we begin the trial there is an easier-to-use diet-tracking program more tailored to the very low-carbohydrate diet, we will consider using that program instead.
- b) Body weight self-monitoring using a digital scale. We will ask participants to track their body weight with an easy-to-use remote scale provided by the study. The scale connects via its own cellular network and therefore does not require any Wi-Fi passwords or setup by participants, simplifying ease of use. We will use this information to monitor participant success and tailor coaching support.
- c) Goals for physical activity and sleep. We will describe the health benefits of physical activity [25]. Using the Diabetes Prevention Program [26] as a guide, participants will be encouraged to engage in moderately intense physical activity for at least 150 minutes a week. The intervention will also describe the connection between lack of sleep and weight gain [27], impaired insulin signaling [28], and type 2 diabetes [29]. Participants will be encouraged to practice sleep hygiene and aim for 7-9 hours a night of sleep.
- d) Training in positive affect and mindfulness (extra psychological supports). We will teach these skills, how they are expected to help, research supporting them, and suggestions for practicing them.
- e) Text messages. Reminders about targeted behaviors are tied to greater behavioral adherence [30, 31]. Thus, to deliver convenient reminders, as Dr. Saslow has done in her previous research, we will send automatic, motivational, and educational skill-relevant messages about 5 times a week to participants [32, 33].
- **f) Mailed materials.** To attempt to help participants change their diet and increase their self-efficacy for new foods, at baseline participants will receive an assortment of difficult-to-find foods that are allowed on their diet (such as coconut and almond flour) and at baseline and 1 and 3 months later we will mail them lay-press cookbooks. Possible materials are pictured to the right.
- **g) Menus**, including written meal plans and grocery lists, will be provided, as these have been found to be more effective for weight loss than an intervention without such support [34].
- h) Access to intervention coach. Coaches have generally been found to be effective additions to behavioral interventions [35]. If participants have questions, they will be able to e-mail their coach whenever they would like in order to receive prompt replies. Phone-based support will also be available on request. We have used this approach successfully in three other online trials of this program for adults with type 2 diabetes. For example, we have a coaching manual that the coach can refer to for common issues. All written coaching messages are vetted by Dr. Saslow before they are sent.
- i) Social support. We will encourage participants to join already existing online, well-moderated support groups for people following an LCD, especially groups for women with PCOS, such as one of the many Facebook or reddit groups. (We will provide a list.) We decided to refer participants to existing groups to ensure long-term access to the groups, a realistic and cost-effective way to provide an intervention at scale.

**Participant safety.** To be responsive to intervention-related health issues that may arise, as in our previous research, we will also inquire about physical symptoms in each weekly e-mail. We will consult with and refer to the participants' primary care physicians as needed. Although we are excluding potential participants with type 1 or 2 diabetes, it is worth noting that diabetic ketoacidosis is a life-threatening complication of poorly controlled diabetes. An LCD reduces the risk of diabetic ketoacidosis; the level of ketones expected in an LCD is an order of magnitude lower than the level seen in diabetic ketoacidosis, and this low level of ketones does not pose a threat to health [36].

To cope with blood pressure changes (as such an approach tends to lower blood pressure), we will teach participants about the signs of low blood pressure, how to self-manage symptoms, and when symptoms may warrant reaching out to their primary care physician for possible medication management.

## 4.0 Statistical Design:

**Power considerations.** As an exploratory study designed to help us understand feasibility and potential efficacy, this trial is not meant to be adequately powered for testing hypothesized effects. Rather it will help us understand the potential efficacy for weight loss and our benchmarks for feasibility (retention, adherence, satisfaction) and other secondary outcomes.

**Data analytic plan.** As we have no control group, we will simply examine means and standard deviations of changes and whether we have reached our benchmarks for the trial. See below for details.

## Intervention outcomes at 4 months

| Intervention feasibility and acceptability | |
|---|---|
| Outcome | Measure/Method |
| Recruitment and retention | We will report numbers for recruitment and retention using a CONSORT diagram. Number and reasons for failure to complete follow-up assessments will be reported. |
| Intervention acceptability and satisfaction | At completion, participants will report the following: 1) satisfaction with each intervention component; 2) satisfaction with the intervention overall; 3) likelihood of referring the intervention to a friend; 4) intervention aspects perceived to be most useful; and 5) suggestions for improvement the intervention. |
| Intervention engagement | Frequency of lesson log-ins and adherence to the recommended diet based on dietary recall. In our previous study in adults with type 2 diabetes, by 4 months participants had logged into more than 95% of lessons. |
| Open-ended questions | We will ask participants open-ended questions about various aspects of their experience to explore, in an open-ended way, their opinion about the intervention and trial. |
| Preliminary efficacy | |
| Primary outcome | Body weight, as measured by a scale we will mail participant (which connects using its own cellular network to our study databases). We will examine the average percent weight loss as well as the percentage of participants in each group who lose a clinically significant amount of weight, at least 5%, which is thought to lead to metabolic improvements and reductions in the future risk of type 2 diabetes [10]. |
| Exploratory metabolic and cardiovascular health outcomes | To reduce the future risk of type 2 diabetes, our goal is to improve glycemic control (glycated hemoglobin; HbA1c), insulin resistance (homeostatic model assessment from fasting blood glucose and insulin; HOMA), lipids (triglycerides and cholesterol), free testosterone [37], and inflammation (C-reactive protein) [38, 39]. These measurements will all occur at MLabs, a local laboratory run by Michigan Medicine. |

### Intervention outcomes at 4 months

| Intervention feasibility and acceptability | |
|---|---|
| Other measures | PCOS-related quality of life [40], general quality of life (from Patient-Reported Outcomes Measurement Information System or PROMIS, which includes depressive symptoms, energy levels, pain, and sleep quality)[41], physical activity [42, 43], dietary adherence (macronutrient levels assessed with a 3-day food record), food cravings [44], stress eating [45, 46], dietary-based social support [47]. |

### References

- 1. Trikudanathan, S., *Polycystic Ovarian Syndrome*. Medical Clinics of North America, 2015. **99**(1): p. 221-235.
- 2. Rotterdam, E. and P. ASRM-Sponsored, *Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS).* Human reproduction (Oxford, England), 2004. **19**(1): p. 41.
- 3. Sam, S., Obesity and Polycystic Ovary Syndrome. Obesity management, 2007. **3**(2): p. 69-73.
- 4. Lim, S.S., et al., *The effect of obesity on polycystic ovary syndrome: a systematic review and meta-analysis.* Obes Rev, 2013. **14**(2): p. 95-109.
- 5. Ezeh, U., B.O. Yildiz, and R. Azziz, *Referral Bias in Defining the Phenotype and Prevalence of Obesity in Polycystic Ovary Syndrome.* The Journal of Clinical Endocrinology and Metabolism, 2013. **98**(6): p. E1088-E1096.
- 6. Yildiz, B.O., E.S. Knochenhauer, and R. Azziz, *Impact of obesity on the risk for polycystic ovary syndrome*. J Clin Endocrinol Metab, 2008. **93**(1): p. 162-8.
- 7. Moran, L.J., et al., *Treatment of obesity in polycystic ovary syndrome: a position statement of the Androgen Excess and Polycystic Ovary Syndrome Society.* Fertility and sterility, 2009. **92**(6): p. 1966-1982.
- 8. Wild, R.A., et al., Assessment of cardiovascular risk and prevention of cardiovascular disease in women with the polycystic ovary syndrome: a consensus statement by the Androgen Excess and Polycystic Ovary Syndrome (AE-PCOS) Society. The Journal of Clinical Endocrinology & Metabolism, 2010. **95**(5): p. 2038-2049.
- 9. Legro, R.S., et al., *Diagnosis and treatment of polycystic ovary syndrome: an Endocrine Society clinical practice guideline.* The Journal of Clinical Endocrinology & Metabolism, 2013. **98**(12): p. 4565-4592.
- 10. Ryan, D.H. and S.R. Yockey, Weight Loss and Improvement in Comorbidity: Differences at 5%, 10%, 15%, and Over. Current Obesity Reports, 2017. **6**(2): p. 187-194.
- 11. Crosignani, P.G., et al., Overweight and obese anovulatory patients with polycystic ovaries: parallel improvements in anthropometric indices, ovarian physiology and fertility rate induced by diet. Hum Reprod, 2003. **18**(9): p. 1928-32.
- 12. Faghfoori, Z., et al., *Nutritional management in women with polycystic ovary syndrome: A review study.*Diabetes & Metabolic Syndrome: Clinical Research & Reviews.
- 13. Thomson, R., J. Buckley, and G. Brinkworth, *Exercise for the treatment and management of overweight women with polycystic ovary syndrome: a review of the literature.* Obesity Reviews, 2011. **12**(5): p. e202-e210.
- 14. Conte, F., et al., *Mental health and physical activity in women with polycystic ovary syndrome: a brief review.* Sports Medicine, 2015. **45**(4): p. 497-504.
- 15. Moran, L.J., et al., *Dietary composition in the treatment of polycystic ovary syndrome: a systematic review to inform evidence-based guidelines.* Journal of the Academy of Nutrition and Dietetics, 2013. **113**(4): p. 520-545.
- 16. Nestler, J.E., et al., Strategies for the use of insulin-sensitizing drugs to treat infertility in women with polycystic ovary syndrome. Fertil Steril, 2002. **77**(2): p. 209-15.

- 17. Legro, R.S., et al., *Prevalence and predictors of risk for type 2 diabetes mellitus and impaired glucose tolerance in polycystic ovary syndrome: a prospective, controlled study in 254 affected women.* Journal of Clinical Endocrinology & Metabolism, 1999. **84**(1): p. 165-169.
- 18. Dunaif, A., *Insulin resistance and the polycystic ovary syndrome: mechanism and implications for pathogenesis.* Endocrine reviews, 1997. **18**(6): p. 774-800.
- 19. Nestler, J.E. and D.J. Jakubowicz, *Decreases in Ovarian Cytochrome P450c17 alpha Activity and Serum Free Testosterone After Reduction of Insulin Secretion in Polycystic Ovary Syndrome.*Obstetrical & gynecological survey, 1997. **52**(2): p. 112-114.
- 20. Gower, B.A., et al., *Favourable metabolic effects of a eucaloric lower-carbohydrate diet in women with PCOS.* Clinical endocrinology, 2013.
- 21. Mavropoulos, J.C., et al., *The effects of a low-carbohydrate, ketogenic diet on the polycystic ovary syndrome: a pilot study.* Nutr Metab (Lond), 2005. **2**: p. 35.
- 22. Saslow, L.R., et al., A randomized pilot trial of a moderate carbohydrate diet compared to a very low carbohydrate diet in overweight or obese individuals with type 2 diabetes mellitus or prediabetes. PLoS One, 2014. **9**(4): p. e91027.
- 23. Saslow, R.L., et al., An Online Intervention Comparing a Very Low-Carbohydrate Ketogenic Diet and Lifestyle Recommendations Versus a Plate Method Diet in Overweight Individuals With Type 2 Diabetes: A Randomized Controlled Trial. J Med Internet Res, 2017. **19**(2): p. e36.
- 24. Trumbo, P., et al., *Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids.* Journal of the American Dietetic Association, 2002. **102**(11): p. 1621.
- 25. Warburton, D.E., C.W. Nicol, and S.S. Bredin, *Health benefits of physical activity: the evidence.* Canadian medical association journal, 2006. **174**(6): p. 801-809.
- 26. Orchard, T.J., et al., *The effect of metformin and intensive lifestyle intervention on the metabolic syndrome: the Diabetes Prevention Program randomized trial.* Annals of Internal Medicine, 2005. **142**(8): p. 611.
- 27. Markwald, R.R., et al., *Impact of insufficient sleep on total daily energy expenditure, food intake, and weight gain.* Proceedings of the National Academy of Sciences, 2013.
- 28. Broussard, J.L., et al., *Impaired Insulin Signaling in Human Adipocytes After Experimental Sleep RestrictionA Randomized, Crossover Study.* Annals of Internal Medicine, 2012. **157**(8): p. 549-557.
- 29. Spiegel, K., et al., *Sleep loss: a novel risk factor for insulin resistance and Type 2 diabetes.* Journal of applied physiology, 2005. **99**(5): p. 2008-2019.
- 30. Fry, J.P. and R.A. Neff, *Periodic prompts and reminders in health promotion and health behavior interventions: systematic review.* Journal of medical Internet research, 2009. **11**(2).
- 31. Pop-Eleches, C., et al., *Mobile Phone Technologies Improve Adherence to Antiretroviral Treatment in Resource-Limited Settings: A Randomized Controlled Trial of Text Message Reminders.* AIDS, 2011. **25**: p. 825-834.
- 32. Chow, C.K., et al., Effect of Lifestyle-Focused Text Messaging on Risk Factor Modification in Patients With Coronary Heart Disease: A Randomized Clinical Trial. JAMA, 2015. **314**(12): p. 1255-1263.
- 33. Redfern, J., et al., *Development of a set of mobile phone text messages designed for prevention of recurrent cardiovascular events.* European journal of preventive cardiology, 2014. **21**(4): p. 492-499.
- 34. Wing, R.R. and R.W. Jeffery, *Food provision as a strategy to promote weight loss.* Obesity research, 2001. **9**(S11): p. 271S-275S.
- 35. Kivelä, K., et al., *The effects of health coaching on adult patients with chronic diseases: A systematic review.* Patient education and counseling, 2014. **97**(2): p. 147-157.
- 36. Phinney, S.D. and J.S. Volek, *The Art and Science of Low Carbohydrate Living: An Expert Guide to Making the Life-saving Benefits of Carbohydrate Restriction Sustainable and Enjoyable*. 2011: Beyond Obesity.
- 37. Lerchbaum, E., et al., *Hyperandrogenemia in polycystic ovary syndrome: exploration of the role of free testosterone and androstenedione in metabolic phenotype.* PLoS One, 2014. **9**(10): p. e108263.
- 38. Gonzalez, F., et al., *Hyperglycemia alters tumor necrosis factor-alpha release from mononuclear cells in women with polycystic ovary syndrome.* J Clin Endocrinol Metab, 2005. **90**(9): p. 5336-42.
- 39. Gonzalez, F., et al., *In vitro evidence that hyperglycemia stimulates tumor necrosis factor-alpha release in obese women with polycystic ovary syndrome.* J Endocrinol, 2006. **188**(3): p. 521-9.

- 40. Cronin, L., et al., *Development of a Health-Related Quality-of-Life Questionnaire (PCOSQ) for Women with Polycystic Ovary Syndrome (PCOS) 1.* Journal of Clinical Endocrinology & Metabolism, 1998. **83**(6): p. 1976-1987.
- 41. Reeve, B.B., et al., Psychometric evaluation and calibration of health-related quality of life item banks: plans for the Patient-Reported Outcomes Measurement Information System (PROMIS). Medical care, 2007. **45**(5): p. S22-S31.
- 42. Craig, C.L., et al., *International physical activity questionnaire: 12-country reliability and validity.* Medicine & Science in Sports & Exercise, 2003. **35**(8): p. 1381-1395.
- 43. Kiernan, M., et al., *The Stanford Leisure-Time Activity Categorical Item (L-Cat): a single categorical item sensitive to physical activity changes in overweight/obese women.* International journal of obesity (2005), 2013. **37**(12): p. 1597.
- 44. Dalton, M., et al., *Preliminary validation and principal components analysis of the Control of Eating Questionnaire (CoEQ) for the experience of food craving.* European journal of clinical nutrition, 2015. **69**(12): p. 1313.
- 45. Tsenkova, V., J.M. Boylan, and C. Ryff, *Stress eating and health. Findings from MIDUS, a national study of US adults.* Appetite, 2013. **69**: p. 151-155.
- 46. Burgess, E., et al., *Profiling motives behind hedonic eating. Preliminary validation of the Palatable Eating Motives Scale.* Appetite, 2014. **72**: p. 66-72.
- 47. Norman, G.J., et al., *Reliability and validity of brief psychosocial measures related to dietary behaviors.* International Journal of Behavioral Nutrition and Physical Activity, 2010. **7**(1): p. 56.